CLINICAL TRIAL: NCT02944565
Title: Daratumumab Infusion Acceleration
Brief Title: Daratumumab in Treating Patients With Multiple Myeloma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OSU-16199; NCI-2016-01504 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2016-10-24; First posted 2016-10-26 (Estimated); Results first posted 2019-09-09 (Actual); Last update posted 2019-09-09 (Actual); Status verified 2019-08

CONDITIONS: Plasma Cell Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — daratumumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (daratumumab) (Experimental): Patients receive daratumumab IV over 1.5 hours. Treatment continues in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Daratumumab

INTERVENTIONS:
Biological: Daratumumab — Given IV
  Other Names: Anti-CD38 Monoclonal Antibody; Darzalex; HuMax-CD38; JNJ-54767414

SUMMARY:
This phase II trial studies the side effects and how well daratumumab works in treating patients with multiple myeloma when the infusion is accelerated. Monoclonal antibodies, such as daratumumab, may interfere with the ability of tumor cells to grow and spread.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the safety and tolerability of decreasing the infusion time of daratumumab in patients that have already received 2+ doses of daratumumab and are continuing on daratumumab.

II. Estimate the time savings versus (vs) predicted infusion time.

OUTLINE:

Patients receive daratumumab intravenously (IV) over 1.5 hours. Treatment continues in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up for 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have received >= 2 daratumumab infusions and be scheduled to receive another dose
* All races and ethnic groups are eligible for this study
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Any other medical condition, including mental illness or substance abuse, deemed by the principal investigator to likely interfere with a patient's ability to sign informed consent, cooperate and participate in the study, or interfere with the interpretation of the results
* Concurrent use of complementary or alternative medicines that in the opinion of the principal investigator would confound the interpretation of toxicities and/or antitumor activity of the study drug
* Prisoner

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2017-02-22 (Actual); Primary Completion 2017-07-20 (Actual); Study Completion 2017-07-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Craig Hofmeister, MD, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (1):
- Ohio State University Comprehensive Cancer Center, Columbus, Ohio, United States

REFERENCES:
- See also: Jamesline — http://cancer.osu.edu

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were enrolled beginning in February 2017 and patient enrollment was completed in June 2017
Groups:
- Treatment (Daratumumab): Patients received daratumumab 16 mg/kg IV over 1.5 hours. Treatment continues in the absence of disease progression or unacceptable toxicity.
Period: Overall Study
Arm/Group | Treatment (Daratumumab)
Started | 28
Completed | 28
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Daratumumab)
Number analyzed (Participants) | 28
Age, Continuous [Median (Full Range); unit: years] | 67 [44 to 90]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 19
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 24
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: patients]
  United States | 28

OUTCOME MEASURES:

1. Primary Outcome: Total Daratumumab Infusion Time
Description: The start and stop times of daratumumab infusion will be tracked during infusion acceleration.
Time Frame: Up to 6 months
Measure: Median (Full Range); unit: hours
Arm/Group | Treatment (Daratumumab)
Number analyzed (Participants) | 28
hours | 1.5 [1.5 to 2.4]

2. Secondary Outcome: Incidence of Adverse Events Defined as Grade 3-4 Reactions Assessed by Common Terminology Criteria for Adverse Events (CTCAE)
Description: Analysis of AEs possibly, probably, or definitely related to protocol therapy will summarize infusion related grade 3-4 reactions.
Time Frame: Up to 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Daratumumab)
Number analyzed (Participants) | 28
Participants | 0

3. Secondary Outcome: Infusion-related Reactions (IRR)
Description: IRR will be assessed during the first infusion using the accelerated dosing regimen. Number of patients who develop grade 3 or above IRR utilizing the accelerated infusion will be used for safety analysis.
Time Frame: Up to 6 months
Measure: Number; unit: participants with IRR
Arm/Group | Treatment (Daratumumab)
Number analyzed (Participants) | 28
participants with IRR | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected at the day of infusion
Arm/Group | Treatment (Daratumumab)
All-Cause Mortality (participants affected / at risk) | 0/28
Serious Adverse Events (participants affected / at risk) | 0/28
Other Adverse Events (participants affected / at risk) | 0/28

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-02-22): https://cdn.clinicaltrials.gov/large-docs/65/NCT02944565/Prot_SAP_000.pdf